CLINICAL TRIAL: NCT04792320
Title: Therapeutic Impact of Oral Uremic Toxin Absorbent and Probiotics in Chronic Kidney Disease Patients With Peripheral Arterial Disease--- on Gut Microbiota, Circulating Long Noncoding RNA, Metabolome, and Vascular Function
Brief Title: Oral Absorbent and Probiotics in CKD Patients With PAD on Gut Microbiota, IncRNA, Metabolome, and Vascular Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202002127RINC
Record Dates: First submitted 2020-05-19; First posted 2021-03-10 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: CKD; PAD - Peripheral Arterial Disease
Keywords: CKD; PAD - Peripheral Arterial Disease; bamboo charcoal probiotics; LncRNA; microbolomics; metabolomics; probiotics
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Active bamboo charcoal (Experimental): Eligible 120 participants (group I),The other 60 eligible controls (group II) will be also randomized into ABC-treatment (A) or no-treatment (B) with a 1:1 ratio. The participants will receive CharXenPlus 4g particles ( containing ABC 2g) thrice daily for 6 months in subgroups IA and IIA.
  While the patients in subgroups IB and IIB will not receive any ABC. The subgroups IA and IB will be further randomly subdivided into IAa, IAb, IBa, and IBb subsubgroups.
  All the patients will receive probiotics APL-MIX2 (CharXprob) 0.8 g powder once a day in the last 3 months except those in subsubgroups IAb and IBb.
  Interventions: Dietary Supplement: Active bamboo charcoal
- Probiotics (Experimental): Eligible 120 participants (group I),The other 60 eligible controls (group II) will be also randomized into ABC-treatment (A) or no-treatment (B) with a 1:1 ratio. The patients will receive CharXenPlus 4g particles ( containing ABC 2g) thrice daily for 6 months in subgroups IA and IIA.
  While the patients in subgroups IB and IIB will not receive any ABC. The subgroups IA and IB will be further randomly subdivided into IAa, IAb, IBa, and IBb subsubgroups.
  All the patients will receive probiotics APL-MIX2 (CharXprob) 0.8 g powder once a day in the last 3 months except those in subsubgroups IAb and IBb.
  Interventions: Dietary Supplement: probiotics
- Active bamboo charcoal+Probiotics (Experimental): Eligible 120 participants (group I),The other 60 eligible controls (group II) will be also randomized into ABC-treatment (A) or no-treatment (B) with a 1:1 ratio. The patients will receive CharXenPlus 4g particles ( containing ABC 2g) thrice daily for 6 months in subgroups IA and IIA.
  While the patients in subgroups IB and IIB will not receive any ABC. The subgroups IA and IB will be further randomly subdivided into IAa, IAb, IBa, and IBb subsubgroups.
  All the patients will receive probiotics APL-MIX2 (CharXprob) 0.8 g powder once a day in the last 3 months except those in subsubgroups IAb and IBb.
  Interventions: Dietary Supplement: Active bamboo charcoal; Dietary Supplement: probiotics
- No invervention (No Intervention): Eligible 120 participants (group I),The other 60 eligible controls (group II) will be also randomized into ABC-treatment (A) or no-treatment (B) with a 1:1 ratio. The patients will receive CharXenPlus 4g particles ( containing ABC 2g) thrice daily for 6 months in subgroups IA and IIA.
  While the patients in subgroups IB and IIB will not receive any ABC. The subgroups IA and IB will be further randomly subdivided into IAa, IAb, IBa, and IBb subsubgroups.
  All the patients will receive probiotics APL-MIX2 (CharXprob) 0.8 g powder once a day in the last 3 months except those in subsubgroups IAb and IBb.

INTERVENTIONS:
Dietary Supplement: Active bamboo charcoal — 4g particle
  Other Names: CharXenPlus
  Arms: Active bamboo charcoal; Active bamboo charcoal+Probiotics
Dietary Supplement: probiotics — 0.8g powder
  Other Names: Charxprob
  Arms: Active bamboo charcoal+Probiotics; Probiotics

SUMMARY:
Taiwan has more chronic kidney disease (CKD) per capita than anywhere in the world, leading to the highest expense of National Health Insurance. By reviewing previous studies, uremic toxins contribute critically to the detrimental effects of CKD on atherosclerotic peripheral artery disease (PAD). When recognized early and managed appropriately, mortality and complications of the participants with CKD and established PAD can be minimized. It is critical to identify novel biomarkers and mediators, which can help identify those with potential poor outcomes and facilitate the discovery/development of novel therapeutics for the patients with CKD and PAD. The OMICs studies support the theory that gut microbiome is a major contributor to adverse cardiovascular outcomes and progression of CKD. However, successful integration of multi-omics approach remains sparse. There is no report on the impact of gut microbiota on the host circulating long non-coding RNAs (lncRNAs) expression signature, other CAD/PAD potential marker, and the potential link between gut microbiota, circulating lncRNA levels changes and CKD/PAD. Additionally, although numerous studies indicated that probiotics or activated charcoal have benefits for CKD patients, few studies evaluated the effect of coadministration of activated charcoal/probiotics on the patients with CKD/PAD. The mechanisms of therapeutic effect on CKD/PAD patients with coadministration of activated charcoal/probiotics involving the cross talk among host, microbiota and metabolites still remain unclear. Thus, in the present study, investigators aim to develop novel diagnostic/prognostic markers and a new treatment with activated bamboo charcoal (ABC)/probiotics for therapeutic opportunities to prevent cardiovascular complications, amputation and death in CKD patients with established PAD. To identify the diagnostic/prognostic markers, the multi-omics (microbolome and metabolome) and lncRNA will be analyzed. The therapeutic impact of activated bamboo charcoal (ABC)/probiotics with optimal formulation, on the renal/endothelial/vascular function, cardiovascular (CV) outcome and mortality in CKD patients with PAD will be also determined to evaluate its therapeutic opportunities.

DETAILED DESCRIPTION:
Taiwan has more chronic kidney disease (CKD) per capita than anywhere in the world, leading to the highest expense of National Health Insurance. By reviewing previous studies, uremic toxins contribute critically to the detrimental effects of CKD on atherosclerotic peripheral artery disease (PAD). When recognized early and managed appropriately, mortality and complications of the participants with CKD and established PAD can be minimized. It is critical to identify novel biomarkers and mediators, which can help identify those with potential poor outcomes and facilitate the discovery/development of novel therapeutics for the participants with CKD and PAD. The OMICs studies support the theory that gut microbiome is a major contributor to adverse cardiovascular outcomes and progression of CKD. However, successful integration of multi-omics approach remains sparse. There is no report on the impact of gut microbiota on the host circulating long non-coding RNAs (lncRNAs) expression signature, other CAD/PAD potential marker, and the potential link between gut microbiota, circulating lncRNA levels changes and CKD/PAD. Additionally, although numerous studies indicated that probiotics or activated charcoal have benefits for CKD patients, few studies evaluated the effect of coadministration of activated charcoal/probiotics on the participants with CKD/PAD. The mechanisms of therapeutic effect on CKD/PAD patients with coadministration of activated charcoal/probiotics involving the cross talk among host, microbiota and metabolites still remain unclear. Thus, in the present study, investigators aim to develop novel diagnostic/prognostic markers and a new treatment with activated bamboo charcoal (ABC)/probiotics for therapeutic opportunities to prevent cardiovascular complications, amputation and death in CKD patients with established PAD. To identify the diagnostic/prognostic markers, the multi-omics (microbolome and metabolome) and lncRNA will be analyzed. The therapeutic impact of activated bamboo charcoal (ABC)/probiotics with optimal formulation, on the renal/endothelial/vascular function, cardiovascular (CV) outcome and mortality in CKD patients with PAD will be also determined to evaluate its therapeutic opportunities. Additionally, the possible mechanisms including the molecular pathway and the roles of microbiota associated with expression profiles of lncRNA and metabolome linked to adverse CV/limb outcome will be investigation. Through combination of innovative molecular biological techniques with new approaches for clinical research, investigators will develop a novel therapy by updated knowledge of the mechanisms of disease and by improved pharmacological technology for the CKD patients with established PAD. Investigators expect to demonstrate the clinical efficacy of ABC ± probiotics to improve symptoms and outcomes of CKD patients with PAD, and offer a possibility to develop a precision medicine with novel diagnostic/prognostic markers and special ABC/probiotic formula, which will ultimately lead to the improved clinical care and outcomes in this population.

ELIGIBILITY:
Inclusion Criteria:

I. CKD/PAD group Patients (Group I)

1. Age > 20 years old on the day of screening.
2. CKD patients with eGFR 15 < eGFR < 60 ml/min/1.73m2 in a stable status, creatinine elevated less than 0.3 mg/dL in at least 30 days before enrollment.
3. Symptomatic PAD with Rutherford Stage ≥ 2 and ABI ≤ 0.9 (or documented by CT-angio, vascular duplex, etc.). II. non-CKD/PAD group Patients (Group II)

1. Age > 20 years old on the day of screening. 2.With eGFR > 60 ml/min/1.73m2 3.No clinical PAD.

Exclusion Criteria:

1. Baseline estimated glomerular filtration rates (eGFR) < 15 ml/min/1.73m2 according to MDRD equation.
2. Patients in severe malnutrition status, albumin less than 2.0 g/dL
3. Patients in severe anemia or active gastrointestinal bleeding with hemoglobulin < 8 g/dL.
4. Peptic ulcer, esophageal varices, ileus or under fasting status
5. Previous gastrointestinal operation.
6. Chronic constipation, as defined with less than 3 bowel movements per week, straining, hard stools, incomplete evacuation and inability to pass stool. If usage of oral laxatives can achieve bowel movement, this patient will not be excluded.
7. Patients with major hemorrhage, as defined with acute hemorrhage and requirement of blood transfusion during index admission.
8. Patients with a biopsy proved or clinically diagnosed advanced liver cirrhosis, Child classification B or C.
9. Solid organ or hematological transplantation recipients.
10. Patients with oliguric kidney injury, as defined with less than 500 cc/day.
11. Evidence of obstructive kidney injury or polycystic kidney disease.
12. Antibiotics or probiotics treatment within the last 2 weeks before enrollment and during follow-up period.
13. Presence or history of malignant neoplasms within the past 5 years prior to the day of screening.
14. Patients with Acquired Immune Deficiency Syndrome.
15. Patients with recent acute coronary syndrome, acute myocardial infarction, or severe heart failure.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-06-19 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
The change of 6-minute walking distance | baseline, 3rd month, 6th month, 1st year, 2nd year and 3rd year
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
The change of ABI | baseline, 3rd month, 6th month, 1st year, 2nd year and 3rd year
  The ABI value is determined by taking the higher pressure of the 2 arteries at the ankle, divided by the brachial arterial systolic pressure.
The change of vascular duplex | baseline, 3rd month, 6th month, 1st year, 2nd year and 3rd year
  Duplex ultrasound of peripheral artery
The change of serum lncRNA | baseline, 3rd month, 6th month, 1st year, 2nd year and 3rd year
  Long non-coding RNAs (long ncRNAs, lncRNA) are a type of RNA, defined as being transcripts with lengths exceeding 200 nucleotides that are not translated into protein.

CONTACTS AND LOCATIONS:
Overall Officials: Chau chung Wu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- NTUH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No